CLINICAL TRIAL: NCT00092404
Title: A Comparison of the Safety, Tolerability, and Immunogenicity of V205C Manufactured With Recombinant Human Albumin (rHA) Versus V205C Manufactured With Pooled-Donor Human Serum Albumin (HSA) in Healthy Children 12 to 18 Months of Age
Brief Title: Safety, Tolerability, and Immunogenicity of an Investigational Vaccine With Recombinant Human Albumin (rHA) in Children 12 to 18 Months of Age (V205C-009)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V205C-009; 2004_074
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — Measles-Mumps-Rubella Vaccine; Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Biological: measles, mumps, and rubella virus vaccine live
  Other Names: V205C
Biological: Comparator: Measles, Mumps, and Rubella Virus Vaccine Live

SUMMARY:
The purpose of this trial is to study the safety and immune response to measles, mumps, and rubella in children who were vaccinated with an investigational measles-mumps-rubella live vaccine made with artificially made human protein.

DETAILED DESCRIPTION:
The duration of treatment is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 12 to 18 months of age

Exclusion Criteria:

* History or prior exposure to measles, mumps, or rubella
* History of allergic reactions to any component of the vaccines as evaluated by the study doctor

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1210 (Actual)
Dates: Start 2001-12; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Antibody response rates to measles, mumps, and rubella at 6 weeks postvaccination | 6 weeks postvaccination

SECONDARY OUTCOMES:
Geometric mean titers to measles, mumps, and rubella by ELISA at 6 weeks postvaccination | 6 weeks postvaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Wiedmann RT, Reisinger KS, Hartzel J, Malacaman E, Senders SD, Giacoletti KE, Shaw E, Kuter BJ, Schodel F, Musey LK. M-M-R((R))II manufactured using recombinant human albumin (rHA) and M-M-R((R))II manufactured using human serum albumin (HSA) exhibit similar safety and immunogenicity profiles when administered as a 2-dose regimen to healthy children. Vaccine. 2015 Apr 27;33(18):2132-40. doi: 10.1016/j.vaccine.2015.03.017. Epub 2015 Mar 18. PMID 25796337
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html